CLINICAL TRIAL: NCT01203878
Title: An Exploratory, Open-label Study of Sequential Field-directed Treatment of Actinic Keratoses of the Face With Imiquimod 3.75% Cream Followed by Photodynamic Therapy
Brief Title: Treatment of Actinic Keratoses of the Face With Imiquimod 3.75% Cream Followed by Photodynamic Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to reach target enrollment of 60 subjects
Sponsor: Tennessee Clinical Research Center (Other)
Collaborators: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09US05N375-Gold
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Actinic Keratosis
Keywords: Imiquimod; Photodynamic therapy; Actinic keratoses; Sequential therapy; Therapeutic uses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy; Aminolevulinic Acid; Solutions; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imiquimod & photodynamic therapy (Experimental): Imiquimod 3.75% applied to the entire face daily for 2 2-week cycles separated by a 2-week no treatment period, followed by one session of photodynamic therapy of the entire face with aminolevulinic acid and blue light
  Interventions: Drug: Photodynamic therapy; Drug: Imiquimod
- Imiquimod (Active Comparator): Imiquimod 3.75% applied to the entire face daily for 2 2-week cycles separated by a 2-week no treatment period, followed by observation
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Photodynamic therapy — Administered 4 weeks after completion of imiquimod therapy
  Other Names: Levulan Kerasticks (aminolevulinic acid 20% solution)
  Arms: Imiquimod & photodynamic therapy
Drug: Imiquimod — Imiquimod 3.75% cream, up to 2 packets, applied topically daily for two 2-week cycles separated by a no-treatment interval of 2-weeks, followed observation
  Other Names: Zyclara (imiquimod 3.75% cream)

SUMMARY:
The purpose of this study is to explore the effect of treating actinic keratoses of the face with imiquimod 3.75% cream followed by photodynamic therapy in comparison to treatment with imiquimod alone

DETAILED DESCRIPTION:
Actinic keratoses are common skin lesions associated with solar ultraviolet radiation exposure. Some actinic keratoses may develop into skin cancers.

Imiquimod 3.75% cream is an approved treatment for actinic keratoses that utilizes a regimen of application to the entire face or balding scalp of up to 2 packets of cream daily for two 2-week cycles, separated by a 2-week no treatment interval.

Photodynamic therapy with aminolevulinic acid (ALA) 20% topical solution is also an approved treatment for actinic keratoses. ALA is applied to actinic keratoses, and after an incubation period, is excited with light. Although approved as a lesion-directed treatment for actinic keratoses, treatment of a field (e.g. face) with photodynamic therapy is commonly performed.

Treatment with photodynamic therapy followed by imiquimod 5% cream has been reported in patients with actinic keratoses, basal cell carcinoma and Bowen's disease, and treatment with imiquimod 5% cream followed by photodynamic therapy in patients with vulvar intraepithelial neoplasia. There are, however, no prior studies on the safety and/or efficacy of using topical imiquimod 3.75% in conjunction with photodynamic therapy in the treatment of actinic keratoses.

This study will use an open-label parallel cohort design in which all patients will received treatment with imiquimod 3.75% cream, and subsequently will be randomized to either photodynamic therapy or observation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults; 18 and over
* At least 10 and no more than 30 clinically typical actinic keratoses on the face

Exclusion Criteria:

* Hypertrophic actinic keratoses or other skin lesions on the head that might required excluded treatment during the study
* Known contraindication to treatment with imiquimod or photodynamic therapy
* Condition that would limit compliance, be a potential safety risk, or require therapy with an excluded treatment
* Systemically immunocompromised
* Pregnant or nursing
* Dermatologic disease and/or condition in treatment area that might exacerbated by treatment with imiquimod, cause difficulty with examination, or require therapy with an excluded treatment
* Participation in another clinical study
* Treatment within the past 60 days with:

  * Ultraviolet therapy
  * Systemic immunomodulators
  * Chemotherapeutic or cytotoxic agents
  * Investigational agents
* Treatment on the head within the past 60 days with:

  * Imiquimod
  * Photodynamic therapy
  * Red or blue light source therapy
  * Cryotherapy or chemotherapy
  * Surgical excision or curettage
  * Topical corticosteroids
  * Laser
  * Dermabrasion
  * Chemical peel
  * Topical retinoids
  * Topical 5-fluorouracil
  * Topical pimecrolimus or tacrolimus
  * Topical diclofenac
* Treatment for actinic keratoses on the head within the past 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, MD, Study Chair — Tennessee Clinical Research Center; Joel Cohen, MD, Principal Investigator — AboutSkin Dermatology and DermSurgery, PC; Girish Munavalli, MD, Principal Investigator — Dermatology, Laser & Vein Specialists of the Carolinas
Locations (3):
- United States (3):
  - AboutSkin Dermatology and DermSurgery, PC, Englewood, Colorado
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from practices of 3 dermatology clinics. First patient enrolled Nov 2010; last patient completed Dec 2011.
Pre-assignment Details: Patients required to complete topical treatment phase prior to randomization to photodynamic therapy or observation. Three subjects discontinued prior to randomization, 2 for adverse events and 1 for withdrawal of consent.
Groups:
- Imiquimod Followed by Photodynamic Therapy: Imiquimod 3.75% applied to the entire face daily for 2 2-week cycles separated by a 2-week no treatment period, followed by one session of photodynamic therapy of the entire face with aminolevulinic acid and blue light
- Imiquimod Followed by Observation: Imiquimod 3.75% applied to the entire face daily for 2 2-week cycles separated by a 2-week no treatment period, followed by observation
- Non-randomized: Imiquimod 3.75% applied to the entire face daily for up to 2 2-week cycles separated by a 2-week no treatment period
Period: Overall Study
Arm/Group | Imiquimod Followed by Photodynamic Therapy | Imiquimod Followed by Observation | Non-randomized
Started | 9 | 9 | 3
Completed | 9 | 9 | 0
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Patients completing week 18 visit
Groups:
- Non-Randomized: Imiquimod 3.75% applied to the entire face daily for up to 2 2-week cycles separated by a 2-week no treatment period,
- Total: Total of all reporting groups
Arm/Group | Imiquimod Followed by Photodynamic Therapy | Imiquimod Followed by Observation | Non-Randomized | Total
Number analyzed (Participants) | 9 | 9 | 3 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 2 | 14
  >=65 years | 3 | 3 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (7) | 61 (6) | 66 (11) | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 7
  Male | 6 | 6 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 3 | 21
Total facial actinic keratosis count [Mean (Standard Deviation); unit: Patient facial actinic keratosis count] | 18.3 (5.6) | 19.9 (5.6) | 18.0 (2.6) | 19.0 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Actinic Keratosis Count
Description: The percent change in actinic keratosis count as compared to the baseline lesion count
Time Frame: Week 18 (4 weeks after randomization visit)
Population: Randomized patients with both a baseline and a week 18 actinic keratosis count. One patient in imiquimod/observation group did not have a baseline count and therefore was not included in the analysis.
Measure: Mean (Standard Deviation); unit: percent reduction in baseline count
Arm/Group | Imiquimod Followed by Photodynamic Therapy | Imiquimod Followed by Observation
Number analyzed (Participants) | 9 | 8
percent reduction in baseline count | 81 (19) | 83 (34)

2. Secondary Outcome: Complete Clearance
Description: The proportion of randomized patients with complete clearance of actinic keratoses in the treatment area (entire face).
Time Frame: Week 18 (4 weeks after randomization visit)
Population: Randomized patients with a week 18 actinic keratosis count.
Measure: Number; unit: participants
Arm/Group | Imiquimod Followed by Photodynamic Therapy | Imiquimod Followed by Observation
Number analyzed (Participants) | 9 | 9
participants | 5 | 2

3. Secondary Outcome: Cosmetic Appearance
Description: Change (improvement) in investigator scores of cosmetic appearance of the treatment area (entire face) by objective and subjective assessments:
  INVESTIGATOR COSMETIC ASSESSMENT 0 - Facial skin is smooth to the touch, without significant lines or unevenness in pigmentation
  1 - Facial skin shows 1 area (cheeks, forehead, or the perioral area) of significant 3 - Facial skin shows 3 areas with significant roughness, dyspigmentation, or fine lines 2 - Facial skin shows 2 areas of significant roughness, dyspigmentation, or fine lines 4 - All are severe in severity
Time Frame: Week 18 (4 weeks after randomization visit)
Population: Randomized patients with both a baseline and a week 18 investigator cosmetic appearance score. One imiquimod/observation patient did not have an end of study investigator cosmetic appearance score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imiquimod Followed by Photodynamic Therapy | Imiquimod Followed by Observation
Number analyzed (Participants) | 9 | 8
units on a scale | 1.67 (1) | 1.25 (0.71)

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: From study entry (Visit 1) to end of study (visit 5).
Arm/Group | Imiquimod Followed by Photodynamic Therapy | Imiquimod Followed by Observation | Non-Randomized
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 5/9 | 4/9 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imiquimod Followed by Photodynamic Therapy (N=9) | Imiquimod Followed by Observation (N=9) | Non-Randomized (N=3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prickly feeling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes labialis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Flu-like symptoms (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fever blister (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Sore on lip (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination (slow enrollment) leading to small numbers of subjects analyzed; missing measurement(s) on a patient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Up to 30 days to review presentations and/or manuscripts. Up to an additional 60 days, if applicable, to file patent applications.